CLINICAL TRIAL: NCT04692142
Title: Comparison Between Different Asynchronous Teaching Methods in an Undergraduate Orthodontic Course: A Crossover Randomised Trial
Brief Title: A Cross-over Randomised Trial Comparing Two Teaching Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PSAU2020030
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Educational Problems
Keywords: Learning; Dental education; Teaching methods; Dental Students

STUDY DESIGN:
Intervention Model Description: The trial is designed as a cross-over clustered randomized trial (each group would be a cluster), so that each group will act as their own control for their learning performance and perception.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor and the statistical analyst will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive online (Active Comparator): Before L1, all students will be asked to complete a set of multiple-choice questions (MCQs), formative exam (i.e. pre-test). Following the test , the lecture will be delivered to the participants of PG using a passive online teaching format for 60 minutes (i.e., live-video streaming). After the lecture is completed, students will be asked to re-take the same pre-test exam and complete questionnaire regarding their experience with the teaching methods.
  Interventions: Other: Flipped classroom teaching method
- Flipped classroom (Experimental): Participants of FG will have an access to a recorded lecture. and they will be taught using an active teaching model known as flipped classroom model. In this model, participants will have 7 -day monitored remote access to the recorded L1. Similar to PG, completing the online pre-test formative exam will be preliminary requirement to access the published recorded L1.
  At the expiry of remote access to the recorded lecture, participants from FG will be invited to attend post-lecture discussion sessions. To enhance the effectiveness of flipped classroom teaching method, the cohort of FG will be randomly, using computer generated randomisation, subdivided to two smaller groups in which each group will be consisted of half of the FG cohort. The same lecturer will moderate the discussions for each group separately. After the lecture is completed, students will be asked to re-take the same pre-test of L1 and complete questionnaire regarding their experience with the teaching methods.
  Interventions: Other: Flipped classroom teaching method

INTERVENTIONS:
Other: Flipped classroom teaching method — Participants will have 7 -day monitored remote access to a recorded lecture about orthodontic topic. At the expiry of remote access to the recorded lecture, participants from FG will be invited to attend post-lecture discussion sessions. To enhance the effectiveness of flipped classroom teaching method, the cohort of FG will be randomly, using computer generated randomisation, subdivided to two smaller groups in which each group will be consisted of half of the FG cohort. The same lecturer will moderate the discussions for each group separately.

SUMMARY:
The aim of the study aim to test the null hypothesis which states that there are no significant differences in knowledge retention and exam performance of dental undergraduate students in a Saudi Dental School using two different asynchronous teaching methods . The secondary aim is to analyse students' perceptions to the two teaching methods.

DETAILED DESCRIPTION:
Design: The trial was designed as a crossover clustered randomized trial whereby each group/ cluster acted as their control for their learning performance and perception.

Setting: College of Dentistry, Princes Sattam Bin Abdulaziz University, Riyadh, Saudi Arabia.

Consents: The ethical approval was obtained from the Scientific Research Unit at the College of Dentistry, Prince Sattam Bin Abdulaziz University, Alkharj, Riyadh (ethical approval PSAU2020030). Written consent was obtained from students before commencing the trial.

Participants: Fourth-year undergraduate dental students enrolled in the preclinical orthodontic course at Prince Sattam University were invited to participate in the study. Students who were registered in the course for the second time were excluded to lessen the bias associated with previous experience of orthodontic teaching. The sample size was based on the total number of students registered in the course at the time of the study.

Randomization: Computer-generated randomization was performed to allocate participants to one of two groups. The sequence of random allocation was concealed from researchers who analyzed the results. Participants in the control group were taught through the virtual traditional learning method (VTL) using live-video streaming, while participants in the intervention group were taught through the virtual flipped learning method (VFL). VTL group included 16 students, while the VFL group included 17 students. We use the term control group to refer to students who studied using the VTL format method across both periods. We also use the term intervention group to refer to students who studied using VFL format across both periods.

Intervention: 4 lectures were delivered asynchronously using two different teaching methods as mentioned above. Participants in VFL had monitored remote access to the recorded lectures for one week, followed by 4 additional small group online discussion sessions. The students in both groups remotely attended all pre-recorded and live-video virtual lectures.

Intervention implementation rounds The intervention was implemented in 3 consecutive weeks. The first lecture (L1: Adult Orthodontics) was taught in the first week. Before L1, all students were asked to complete a set of multiple-choice questions (MCQs) formative exam (i.e., pre-test). Following the pre-test, the lecture was delivered to participants of the VTL group using a passive online teaching format (live-video streaming). L1 was also recorded after obtaining verbal consent from the attendees. After the lecture was completed, students were asked to re-take the same pre-test exam and complete a questionnaire regarding the VTL experience.

Within 24 hours following L1, participants of VFL had 7-day monitored remote access to the recorded lecture of L1, and they were taught using an active teaching model, referred to as the VFL model. Like the participants of the VTL group, participants of the VFL group were asked to complete the relevant pre-test.

At the expiry of remote access to the recorded lecture, participants from VFL were invited to attend post-lecture discussion sessions. To enhance the effectiveness of post-lecture discussion, participants were randomly divided into two smaller subgroups, and the same lecturer facilitated the discussions for each group separately. At the end of each discussion session, participants were asked to re-take the pre-test of L1 and a complete questionnaire regarding their VFL experience.

Following the small group's discussion session, participants of VFL were given a 30-minute break before the start of the second lecture related to the topic of Orthognathic Surgery (L2). However, the intervention was crossed over; hence, the cohort of VFL in week 1 acted as a control group while teaching L2 and vice versa. The same protocol of teaching models that were applied in week 1 was adopted.

Participants of both groups were taught by the same instructor using the same materials, irrespective of the teaching methods. The lectures were delivered using the same presentation platform (PowerPoint, Microsoft Corp, Redmond, WA) and the same virtual learning platform (Zoom live-streaming software - Zoom Video Communications, Inc, San Jose, California, Version 5.4.3). The duration of each lecture was 60 minutes, while the post-lecture discussion in the VFL design lasted 15 minutes. Learning outcomes were based on each lecture's learning objectives and outcomes that aligned with what is specified by the National Commission for Academic Accreditation and Assessment in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* Fourth-year undergraduate students enrolled in the course, in a Saudi Dental college.

Exclusion Criteria:

* Students who are enrolled in the course for a second time

Ages: 22 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The institution where the study will be carried on enrolls only male dental students.
Enrollment: 32 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Formative exam | 7-days
  Before each lecture, students will complete a set of multiple-choice questions (MCQs), formatively (i.e. pre-test). These questions will be related to the taught topics, and will be administered remotely using learning management system (Blackboard). After each lecture, students will be asked to re-take the same pre-test via Blackboard. This formative assessment test will measure students' learning gain. Two investigators will construct the pre-test questions to ensure its content validity and reliability. Content validity will be tested using test matrix and experts judgment. The reliability test will estimated using inter-rater reliability. A correlation of more than 0.7 will be considered acceptable.

SECONDARY OUTCOMES:
Perception to the two teaching methods. | 7-days
  At the end of each lecture, students will be asked to answer a questionnaire regarding their experience with the teaching methods they have received. We will use the validated Web-Based Learning Environment Inventory (WELEI), developed by Chang and Fisher (2001). In addition to demographic section, the questionnaire consists of items that captures students' perceptions of web-based learning environments. Regarding the flipped classroom teaching method, we will include additional questions adapted from previous studies that examined students' perception of the flipped classroom (Johnson, 2013 and Butt, 2014). The questionnaire will be distributed online via SurveyMonkey (San Mateo, California, United States).

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alharbi, PhD, Study Chair — Prince Sattam Bin Abdulaziz University
Locations (1):
- Prince Sattam Bin Abdulaziz University, Al Kharjah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon asking.
Supporting Information: Study Protocol
Time Frame: Within one year
Access Criteria: Eligible researcher who does a similar research.

REFERENCES:
- [Derived] Alharbi F, Alwadei SH, Alwadei A, Asiri S, Alwadei F, Alqerban A, Almuzian M. Comparison between two asynchronous teaching methods in an undergraduate dental course: a pilot study. BMC Med Educ. 2022 Jun 23;22(1):488. doi: 10.1186/s12909-022-03557-7. PMID 35739594